CLINICAL TRIAL: NCT06655428
Title: The REDUCE EU Study - Endobronchial Thermal Liquid Ablation (ETLA) for the Treatment of Emphysema - A Pilot Study (CSP-12123)
Brief Title: The REDUCE EU Study - Endobronchial Thermal Liquid Ablation (ETLA) for the Treatment of Emphysema
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Morair Medtech, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP-12123; CIV-24-04-046660 (Other: European Commission)
Record Dates: First submitted 2024-10-17; First posted 2024-10-23 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Emphysema or COPD; Emphysema; Emphysema, Pulmonary; COPD; COPD (Chronic Obstructive Pulmonary Disease)
Keywords: Lung Volume Reduction; bronchoscopic lung volume reduction; ETLA; BTVA; LVR; Lung Disease, obstructive; Chronic Obstructive Lung Disease; Respiratory Tract Disease
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive; Pulmonary Emphysema; Lung Diseases, Obstructive; Respiratory Tract Diseases | interventions — Pneumonectomy

STUDY DESIGN:
Intervention Model Description: The study is prospective, single-arm and multi-center.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Endobronchial Thermal Liquid Ablation (ETLA) Treatment (Experimental): Participants will undergo up to two ETLA procedures separated by a minimum three-month interval.
  Interventions: Device: Endobronchial Therman Liquid Ablation (ETLA)

INTERVENTIONS:
Device: Endobronchial Therman Liquid Ablation (ETLA) — The ETLA System is a minimally invasive bronchoscopic treatment designed to deliver heated normal saline to targeted emphysematous lung regions with hyperinflation to cause tissue ablation and subsequent volume reduction as a means for treating emphysema. The ETLA procedures will be performed under general anesthesia. Each procedure will be limited to treatment in a single lung, with either unilateral or bilateral treatment over the two procedures.
  Other Names: Bronchoscopic lung volume reduction

SUMMARY:
The goal of this clinical trial is to learn if bronchoscopic lung volume reduction with endobronchial thermal liquid ablation (ETLA) works to treat severe emphysema in terms of feasibility and safety.

Participants will:

* Have up to two ETLA procedures
* Complete five clinic follow-up visits and two virtual follow-up visits.

DETAILED DESCRIPTION:
ETLA offers the potential to result in significant lung volume reduction of hyperinflated emphysematous regions, providing clinically meaningful improvement in pulmonary function and quality of life to a broad population of patients with severe emphysema. The REDUCE EU Pilot study will primarily evaluate the feasibility and safety of ETLA treatment in patients with severe emphysema. Secondarily, the study will evaluate the efficacy of sequential ETLA treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years old
* Diagnosis of COPD with FEV1/FVC less than 0.7 post-bronchodilation
* Post-bronchodilator Forced Expiratory Volume (FEV1) ≥ 20% and ≤ 49% of predicted value
* Total lung capacity (TLC) ≥ 100% predicted
* Residual volume (RV) ≥ 175% predicted
* 6 Minute Walk Distance (6MWD) ≥ 140 meters
* Dyspnea scoring ≥ 1 on the modified Medical Research Council scale (mMRC)
* Blood gas values of PCO2 ≤ 55 mmHg; PO2 ≥ 45 mmHg on room air
* Optimized medical management (consistent with GOLD guidelines) as confirmed by the Investigator
* Non-smoking for 3 months prior to study enrollment, as confirmed by lab testing
* Participant must engages in physical exercise beyond activities of daily living (i.e., a walking program, pulmonary rehabilitation) on n a regular basis for more than 6 weeks prior to enrollment and agree to continue the activity throughout study participation
* Participant must live within approximately 1 hour of the study hospital, or live within 1 hour of adequate regional care, or be willing to remain in the hospital for at least five days post-procedure
* Vaccinated for COVID-19, pneumococcus, and influenza (per European Union and Member State guidelines) or documented clinical intolerance or documented patient refusal
* Cognitively able to provide written informed consent and willing to comply with study requirements
* Severe emphysematous lung subsegments eligible for ETLA treatment

Exclusion Criteria:

* Body mass index (BMI) < 16 kg/m^2 or ≥ 33 kg/m^2
* DLCO < 20% predicted
* Chronic bronchitis as defined by cough and sputum production for at least 3 months per year for two consecutive years, in the absence of other conditions that can explain these symptoms
* 75ml or greater sputum production per day most days of the week
* Greater than two hospitalizations for COPD exacerbations and/or pneumonia in the 12 months prior to enrollment
* Diagnosis of asthma that is confirmed according to the Global Initiative for Asthma (GINA) guidelines
* Prior lung volume reduction via endobronchial valves(s), coil(s), vapor and/or polymer. Patients whose valves have been removed > 3 months previously can be treated if a baseline bronchoscopy reveals no airway obstruction or obvious tissue granulation and the reason for valve removal was not for complications e.g., Pneumonia, severe exacerbation, or pneumothorax.
* Pulmonary hypertension
* Alpha-1 antitrypsin deficiency
* Uncontrolled diabetes mellitus
* Prior heart or lung transplant
* Myocardial infarction or stroke within the 12 months of enrollment
* Diagnosis of heart failure
* Heart failure requiring hospitalization, within 6 months prior to enrollment
* History of bleeding disorders or enhanced predisposition to bleeding
* History of severe/massive hemoptysis defined as >200ml of blood loss in < 24 hours
* Unable to discontinue anti-coagulants or platelet inhibitors (acetylsalicylic acid [ASA]and non-ASA, including low dose) for at least 7 days prior to each procedure (or as per physician discretion based on the specific agent) and for at least 6 weeks after each procedure
* Daily systemic steroids equivalent to > 15mg prednisolone
* Immunosuppressive drugs, such as for the treatment of cancer, autoimmune disease, or prevention of tissue/organ rejection
* Pregnant, lactating, or women of childbearing potential that plan to become pregnant within the study duration
* Currently enrolled in another trial studying an experimental treatment
* Any disease or condition likely to limit survival to less than one year
* Concomitant illnesses or medications that may pose a significant increased risk for complications following treatment with ETLA
* Any condition that would interfere with evaluation or completion of the study including study assessments and procedures, including bronchoscopy.
* Active aspergillus infection
* Clinically significant bronchiectasis as determined by the Investigator
* Radiological evidence of bronchiectasis in target region(s) and/or cystic radiological bronchiectasis in any region of the lungs
* Clinically significant pulmonary fibrosis
* Lung nodule not proven stable unless proven to have benign pathology
* Large bulla (defined as > 1/3 volume of a lung)
* Prior Lung Volume Reduction Surgery (LVRS), bullectomy, or lobectomy
* The remaining lung tissue NOT targeted for ETLA treatment is too highly diseased
* Active respiratory infection or recent respiratory infection with resolution < 4 weeks prior to screening or procedure
* Recent COPD exacerbation within < 6 weeks prior to screening or procedure

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Percent of procedures where the device operated as intended | Through completion of the second procedure, approximately 13 weeks
  Percent of procedures where the device operated as intended per the Instructions for Use (IFU)
Incidence of serious adverse events (SAE) | 6 months
  Incidence of serious adverse events (SAE) associated with the ETLA device and/or procedure as adjudicated by an independent medical monitor.

SECONDARY OUTCOMES:
Incidence of adverse events | 9 months
  Incidence of all adverse events associated with the ETLA device and/or procedure
Incidence of serious adverse events (SAE) | 9 months
  Incidence of serious adverse events (SAE) associated with the ETLA device and/or procedure as adjudicated by an independent medical monitor
Residual volume (RV) change | 3, 6, and 9 months
  Change in residual volume (RV) (mL, % change in absolute and % predicted)
FEV1 change | 3, 6, and 9 months
  Change in Forced Expiratory Volume in the first second (FEV1) (mL, % change in absolute and % predicted)
RV/TLC change | 3, 6, and 9 months
  Change in residual volume (RV) over total lung capacity (TLC) (RV/TLC)
6MWT change | 3, 6, and 9 months
  Change in Six Minute Walk Test (6MWT)
SGRQ-C change | 3, 6, and 9 months
  Change in SGRQ-C (Saint George Respiratory Questionnaire-COPD)

OTHER OUTCOMES:
Target Lobe Volume Reduction | Baseline to 3 months post-procedure 1, 3 months post-procedure 1 to 3 months post-procedure 2
  Target Lobe Volume Reduction (TLVR) as measured by CT scan quantified by the reduction in the volume of the targeted lobe(s) (reported in mL)
Cumulative Lobar Volume Reduction | Through follow-up of the second procedure, approximately 6 Months
  Cumulative Lobar Volume Reduction as measured by CT scan, quantified by the summation of TLVR through both procedures (reported in mL)
Catheter positioning allowing treatment | Through completion of the second procedure, approximately 13 weeks
  Percent of target regions where the catheter is placed in the target airway with positioning allowing treatment
Heated saline at predetermined volume | Through completion of the second procedure, approximately 13 weeks
  Percent of target regions where heated saline is delivered at the predetermined volume per treatment plan
Auxiliary reduction | Through follow-up of the second procedure, approximately 6 Months
  Number of procedures where auxiliary reduction is observed in a region not predicted
Responder analyses | 3, 6, and 9 months
  Responder analyses for:
  * Improvement in FEV1 of ≥ 12%
  * Reduction in RV of ≥ 6%
  * Reduction in RV/TLC of ≥ 3%
  * Increase in 6MWD of ≥ 26 meters
  * Improvement in SGRQ-C of ≥ 4 points
TLC change | 3, 6, and 9 months
  Change in Total Lung Capacity (TLC)
CAT score change | 3, 6, and 9 months
  Change in COPD Assessment Test (CAT) score
BODE index change | 3, 6, and 9 months
  Change in BODE index (body-mass index, airflow obstruction, dyspnea, and exercise)
DLCO change | 3, 6, and 9 months
  Change in DLCO (lung diffusion test)
mMRC change | 3, 6, and 9 months
  Change in mMRC (Modified Medical Research Council dyspnea questionnaire)

CONTACTS AND LOCATIONS:
Locations (7):
- Austria (2):
  - Universitätsklinikum Allgemeines Krankenhaus Wien, Vienna, Austria
  - Klinik Floridsdorf, Vienna, Austria
- Germany (4):
  - Gemeinschaftskrankenhaus Havelhöhe gGmbH Klinik für Anthroposophische Medizin, Berlin, Germany
  - Asklepios Lungenklinik Gauting GmbH, Gauting, Germany
  - Asklepios Klinik Barmbek, Hamburg, Germany
  - Thoraxklinik University of Heidelberg, Heidelberg, Germany
- University Medical Center Groningen, Groningen, The Netherlands, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided